CLINICAL TRIAL: NCT00122499
Title: A Study to Assess the Efficacy of Tadalafil to Treat Erectile Dysfunction After Radiotherapy of Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 232.476/2003/180
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2005-07-27 (Estimated); Status verified 2005-07

CONDITIONS: Prostate Cancer; Erectile Dysfunction
Keywords: Prostate cancer; Radiotherapy; Erectile dysfunction; Tadalafil
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Tadalafil

INTERVENTIONS:
Drug: tadalafil

SUMMARY:
This study has been designed to evaluate the efficacy and safety of a 20-mg dose of tadalafil administered "on demand" to patients with erectile dysfunction (ED) after external-beam radiotherapy (EBRT) of prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer has become the most frequent malignancy in older men in Western countries. Radiotherapy is a common treatment modality for early stage prostate cancer. Because of the high incidence of post-radiation erectile dysfunction (ED), up to 72% after external-beam radiotherapy, this patient category represents a most difficult therapeutic challenge. Oral drug therapy represents the first-line management option for patients with ED. The results of the studies completed thus far with sildenafil show that a phosphodiesterase type 5 inhibitor is a safe and efficacious drug for the treatment of post-radiation ED. No studies have investigated the efficacy of tadalafil in men complaining of ED after radiotherapy of prostate cancer. Because of the extended period of effectiveness, which may last up to 36 hours after intake, tadalafil allows freedom in the choice for time of sexual activity. Also the absence of restrictions of tadalafil intake with food or alcohol should simplify its administration. This randomized, double-blind, placebo-controlled, cross-over study has been designed to evaluate the efficacy and safety of "on demand" dosing of 20-mg of tadalafil or placebo administered for 12 weeks to patients with ED after external-beam radiotherapy for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual men, at least 18 years of age at Visit 1 and willing to participate in the study. If a qualifying participant has more than one female sexual partner during the study, the participant will not be excluded from the trial. However, the participant will be required to respond to the questionnaires based on the participant's sexual interactions with only one of these partners.
* Patients with histologically proven prostate cancer.
* Provide signed informed consent.
* Developed ED (defined as a consistent change in the quality of erection that adversely affects the patient's satisfaction with sexual intercourse) subsequent to EBRT for prostate cancer.
* Patients willing to make on average 1 sexual intercourse attempt every week during the study (including the 4-week run-in period without medication).
* Agree not to use any other ED treatment for at least 4 weeks before receiving the initial dose of study drug (ie, during the run-in period and during the treatment phase of the study).
* Have been treated by EBRT at least 12 months before screening and were documented to be potent before undergoing EBRT.

Exclusion Criteria:

* Patients will not be randomized if they did not make at least 1 sexual intercourse attempt during the run-in period. Also patients who are unable to appropriately complete the questionnaires will not be randomized.
* ED caused by other primary sexual disorders including premature ejaculation or ED caused by untreated endocrine disease (eg, hypopituitarism, hypothyroidism, or hypogonadism).
* History of pelvic surgery (including radical prostatectomy)
* Treatment with cancer chemotherapy or anti-androgens.
* Have a raising prostate specific antigen level or metastases at Visit 1.
* History of penile implant.
* The presence of clinically significant penile deformity in the opinion of the investigator.
* Evidence of clinically significant renal insufficiency within the last 6 months before Visit 1.
* Active symptomatic hepatobiliary disease, including patients with evidence of jaundice at Visit 1.
* Patients with chronic stable angina treated with long-acting nitrates, or patients with chronic stable angina who have required short-acting nitrates in the last 90 days, or angina occurring during sexual intercourse in the last 6 months.
* Patients having met the criteria for unstable angina (Braunwald, 1989) within 6 months before Visit 1, history of myocardial infarction or coronary artery bypass graft surgery within 90 days before Visit 1, or percutaneous coronary intervention (eg, angioplasty or stent placement) within 90 days before Visit 1.
* Any supraventricular arrhythmia with an uncontrolled ventricular response (mean heart rate >100 bpm) at rest despite medical or device therapy, or any history of spontaneous or induced sustained ventricular tachycardia (heart rate >100 bpm for ≥ 30 sec) despite medical or device therapy, or the presence of an automatic internal cardioverter-defibrillator.
* A history of sudden cardiac arrest despite medical or device therapy.
* Any evidence of congestive heart failure class 2 or above within 6 months before Visit 1 (Criteria Committee, New York Heart Association, Inc., 1964).
* A new, significant conduction defect within 90 days before Visit 1.
* Systolic blood pressure >170 or <90 mm Hg or diastolic blood pressure >100 or <50 mm Hg, or patients with a history of malignant hypertension.
* History of significant central nervous system injuries (including stroke and spinal cord injury) within the 6 months before Visit 1.
* History of HIV infection.
* Any condition that would interfere with the patient's ability to provide informed consent or comply with study instructions, would place patient at increased risk, or might confound the interpretation of the study results.
* History of drug, alcohol, or substance abuse within the 6 months before Visit 1.
* Treatment within the 30 days before Visit 1 with a drug or device that has not received regulatory approval.
* Have any condition, limitation, or disease that could, in the judgment of the investigator, preclude evaluation of response to tadalafil.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Study Completion 2005-02

PRIMARY OUTCOMES:
To evaluate the efficacy of 20 mg tadalafil, in comparison with placebo, in men with ED after 3-D conformal radiotherapy (3DCRT) of prostate cancer

SECONDARY OUTCOMES:
Responses to the Global Assessment Questions (GAQ), and the other items of the Sexual Encounter Profile (SEP) and International Index of Erectile Function (IIEF)
To assess the side effects of 20 mg tadalafil in men with ED after 3DCRT

CONTACTS AND LOCATIONS:
Overall Officials: Luca Incrocci, M.D., Ph.D., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands